CLINICAL TRIAL: NCT03997955
Title: Myofascial Induction Effects on Plantar Pressures and Stabilometry Variables. A Clinical Trial
Brief Title: Myofascial Induction Effects on Plantar Pressures and Stabilometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Principal Investigator, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Myofascial-Induction_CT
Record Dates: First submitted 2019-06-23; First posted 2019-06-25 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Foot Diseases; Myofascial Pain
MeSH Terms: conditions — Foot Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Myofascial induction
  Interventions: Other: Myofascial induction
- Control group (Sham Comparator): Sham myofascial induction
  Interventions: Other: Sham myofascial induction

INTERVENTIONS:
Other: Myofascial induction — Myofascial induction in plantar fascia
  Arms: Experimental group
Other: Sham myofascial induction — Sham myofascial induction in plantar fascia
  Arms: Control group

SUMMARY:
The objective is to determine the effectiveness of myofascial Induction effects on plantar pressures and stabilometry variables. Forty healthy subjects (28 females and 12 males) will be recruited for a simple blind clinical trial. All subjects will be randomly distributed in two different groups: control group (sham treatment of myofascial Induction) and experimental group (myofascial Induction). Outcome measurements will be foot plantar pressure area (footprint) and center of pressure area (stabilometry) by the Balance Evaluation Systems test. Two trials will be recorded for each condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without pain.

Exclusion Criteria:

* Previous lower extremities surgery
* History of lower extremities injury with residual symptoms within the last year
* Evidence of a leg-length discrepancy of more than 1 cm
* Evidence of balance deficits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Foot plantar pressure area | Change from foot plantar pressure area at 2 minutes
  Foot plantar pressure area measured by the Balance Evaluation Systems test (squared centimeters)

SECONDARY OUTCOMES:
Center of pressure area | Change from center of pressure area at 2 minutes
  Center of pressure area measured by the Balance Evaluation Systems test (squared centimeters)

CONTACTS AND LOCATIONS:
Locations (1):
- Eva María Martínez, Madrid, Spain

REFERENCES:
- [Derived] Martinez-Jimenez EM, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Diaz-Velazquez JI, Palomo-Lopez P, Rodriguez-Sanz D, Calvo-Lobo C, Lopez-Lopez D. Pressure and Traction Technique Improves Postural Control More Than Tactile Stimulation in Foot Plantar Fascia: A Randomized Single-Blind Trial. Arch Phys Med Rehabil. 2020 Jun;101(6):978-984. doi: 10.1016/j.apmr.2020.01.017. Epub 2020 Feb 28. PMID 32113972